CLINICAL TRIAL: NCT00068887
Title: Regional Fatty Acid Metabolism in Humans
Status: Withdrawn | Type: Observational
Why Stopped: NOT A CLINICAL TRIAL
Sponsor: Mayo Clinic (Other)
Other Study IDs: RFAMH (DK45343) (withdrawn)
Record Dates: First submitted 2003-09-10; First posted 2003-09-12 (Estimated); Last update posted 2015-04-30 (Estimated); Status verified 2015-04

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: type 2 diabetes; some studies - family history of type 2 diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
There are several studies looking at how dietary fat is metabolized by humans. We give special meals and collect blood, breath, urine and fat samples to study how people burn and store dietary fat.

ELIGIBILITY:
Inclusion Criteria: BMI<25 Lean, sedentary with family history of DM2 and Lean, sedentary without family history of DM2 and Lean, active without family history of DM2. Non-smokers.

Exclusion Criteria: Known systemic illness, cardiac and vascular disease and BP> 160/95 on HTN meds. Medications that affect fat metabolism.

We do not pay for travel expenses.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 1999-09; Study Completion 2005-12

CONTACTS AND LOCATIONS:
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States